CLINICAL TRIAL: NCT05173714
Title: Sit Less, Interact and Move More (SLIMM) 2 Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Srinvasan Beddhu (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Stanford University (Other)
Responsible Party: Sponsor-Investigator, Srinvasan Beddhu, Professor, Internal Medicine, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 138494; 1R01DK128640-01 (NIH)
Record Dates: First submitted 2021-11-04; First posted 2021-12-30 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Diseases; Obesity
MeSH Terms: conditions — Renal Insufficiency, Chronic; Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- SLIMM + Standard RT + Placebo (Placebo Comparator): SLIMM intervention for 3 months, followed by a 9-month intervention of SLIMM, standard-of-care resistance training and oral placebo
  Interventions: Behavioral: SLIMM; Behavioral: Standard Resistance Training; Drug: Placebo
- SLIMM + Guided RT + Placebo (Active Comparator): SLIMM intervention for 3 months, followed by a 9-month intervention of SLIMM, guided resistance training and oral placebo
  Interventions: Behavioral: SLIMM; Behavioral: Guided Resistance Training; Drug: Placebo
- SLIMM + Guided RT + Semaglutide (Experimental): SLIMM intervention for 3 months, followed by a 9-month intervention of SLIMM, guided resistance training and oral semaglutide
  Interventions: Behavioral: SLIMM; Behavioral: Guided Resistance Training; Drug: Semaglutide

INTERVENTIONS:
Behavioral: SLIMM — Increase in light walking activity, replacing 1 hour/day of sedentary duration with casual walking duration. Increase in sedentary breaks, from sitting/lying position to standing position, at least once every hour as independent of the total time spent on sedentary activities.
Behavioral: Standard Resistance Training — Participants will be provided a standard resistance training regimen to follow during the course of the study. Participants will not receive individualized instruction, guidance or modification to the resistance training regimen.
  Arms: SLIMM + Standard RT + Placebo
Behavioral: Guided Resistance Training — Supervised resistance training sessions are individualized for a low-resistance, high-repetition regimen of lower body major muscle groups with established guidelines. Instructions and resistance training bands will be provided for home use. Study participants will record compliance to the resistance training regimen for further guidance and potential modification.
  Arms: SLIMM + Guided RT + Placebo; SLIMM + Guided RT + Semaglutide
Drug: Placebo — Oral placebo tablets (matching the experimental semaglutide) will be administered from the first through ninth months of the drug intervention period.
  Arms: SLIMM + Guided RT + Placebo; SLIMM + Standard RT + Placebo
Drug: Semaglutide — Oral semaglutide 3 mg/day will be administered for the first month of study drug intervention period, if tolerated, the dose will increase to 7 mg/day for the second month and to a maximum dose of 14 mg/day from the third through ninth months of the drug intervention period.
  Arms: SLIMM + Guided RT + Semaglutide

SUMMARY:
* Prolonged sitting (sedentary behavior) is a risk factor for decreased kidney function, obesity, diabetes and mortality. Prolonged sitting is associated with decreased kidney function and increased risk of diabetes, heart disease and death.
* In a previous pilot study funded by NIH, it was shown that a Sit Less, Interact and Move More (SLIMM) intervention targeting sedentary behavior in people with kidney disease was able to decrease prolonged sitting but that effect was not sustained.
* Therefore, the researchers are currently conducting a follow-up study named Sit Less, Interact and Move More (SLIMM) 2.
* This NIH funded study is conducted at the University of Utah and Stanford University.
* The purpose of this study is to see if guided resistance training (to improve muscle strength) and semaglutide (FDA approved diabetes and weight loss medication that might also improve physical function) can boost adherence to the SLIMM Intervention and reduce sedentary behavior.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Glomerular Filtration Rate (eGFR) 20 to <60 mL/min/1.73m^2
* Able to perform resistance training
* Access to compatible "smartphone" or device (i.e., Android, Kindle or Apple with internet connectivity or mobile network), desktop or laptop

Exclusion Criteria:

* Type 1 Diabetes
* History of gastroparesis or paralytic ileus
* At baseline, if sedentary time is 25 min/hr or less, measured by accelerometer
* Potential contraindications to semaglutide such as a history of pancreatitis, and a family or personal history of multiple endocrine neoplasia type 2 or familial medullary thyroid carcinoma.
* Previous bariatric surgery
* Medical condition likely to limit survival to less than 1 year
* Anticipated start of dialysis or kidney transplantation within 6 months
* Any factors judged by the investigator or study team to likely limit adherence to interventions
* Vulnerable populations- pregnant or incarcerated
* Enrolled in interventional trials using drugs or devices
* Not able to undergo informed consent
* Recent hospitalizations or major interventional procedures done within the past 60 days
* Known or suspected hypersensitivity to tegaderm
* Use of any GLP-1 receptor agonist within 30 days prior to screening
* Presently classified as being in New York Heart Association (NYHA) Class IV Heart Failure
* Daytime use of supplemental oxygen (i.e., prescribed a stationary or portable oxygen system)
* Presence of metastatic cancer
* Current use of mobility aid(s)
* Living in the same household of a participant already enrolled in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Average Change in Sedentary Duration at Months 8, 10 and 12 from Randomization | Randomization to 12 Months
  The primary analysis will provide estimates and confidence intervals for the three arms comparisons of changes in sedentary duration from randomization (at 3 months) to the average of changes at months 8, 10 and 12 between the randomized groups that constitute the co-primary comparisons under the study design

SECONDARY OUTCOMES:
Average Change in Steps per Day at Months 8, 10 and 12 from Randomization | Randomization to 12 Months
  The analysis will provide estimates and confidence intervals for the three arms comparisons of changes in steps per day from randomization (at 3 months) to the average of changes at months 8, 10 and 12 between the randomized groups.
Average Change in Stepping Duration at Months 8, 10 and 12 from Randomization | Randomization to 12 Months
  The analysis will provide estimates and confidence intervals for the three arms comparisons of changes in stepping duration from randomization (at 3 months) to the average of changes at months 8, 10 and 12 between the randomized groups.
Average Change in Six-Minute Walk at Months 6 and 12 from Randomization | Randomization to 12 Months
  Changes in six minute walk distance from randomization (at 3 months) to the average of changes at months 6 and 12
Average Change in Body Fat % at Months 6 and 12 from Randomization | Randomization to 12 Months
  Changes in average body fat percentage as measured by bioimpedance analysis from randomization (at 3 months) to the average of changes at months 6 and 12

OTHER OUTCOMES:
Average Change in Patient Reported Fatigue at Months 6 and 12 from Randomization | Randomization to 12 Months
  Changes in patient reported fatigue as measured by questionaires from randomization (at 3 months) to the average of changes at months 6 and 12
Average Change in Patient Reported Sleep at Months 6 and 12 from Randomization | Randomization to 12 Months
  Changes in patient reported sleep as measured by questionaires from randomization (at 3 months) to the average of changes at months 6 and 12
Average Change in Patient Reported Quality of Life at Months 6 and 12 from Randomization | Randomization to 12 Months
  Changes in patient reported quality of life as measured by questionaires from randomization (at 3 months) to the average of changes at months 6 and 12
Average Change in Lower Extremity Performance Battery Composite Score (LEP-CS) at Months 6 and 12 from Randomization | Randomization to 12 Months
  Changes in Lower Extremity Performance Battery Composite Score (LEP-CS) from randomization (at 3 months) to the average of changes at months 6 and 12
Average Change in Circulating Protein Markers of Inflammation at Months 6 and 12 from Randomization | Randomization to 12 Months
  Changes in circulating protein markers of inflammation from randomization (at 3 months) to the average of changes at months 6 and 12
Average Change in microRNA (miRNA) Markers of Inflammation at Months 6 and 12 from Randomization | Randomization to 12 Months
  Changes in microRNA (miRNA) markers of inflammation from randomization (at 3 months) to the average of changes at months 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Srinivasan Beddhu, M.D., Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No